CLINICAL TRIAL: NCT00308009
Title: Multicenter Prospective Randomized Trial Comparing to Strategies When Incontinence Surgery is Needed in Addition to Prolapse Surgery
Brief Title: Comparison of the Result of TVT Performed at the Time of Prolapse Surgery or 3 Months After
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Ellen Borstad, MD, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVT Prolapse study
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2007-11

CONDITIONS: Pelvic Organ Prolapse; Urinary Stress Incontinence
Keywords: Pelvic Organ Prolapse; Urinary stress incontinence; Surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Group I, Prolapse repair and TVT concomitantly
  Interventions: Procedure: Vaginal Repair for prolapse, TVT procedure; Procedure: TVT and Prolapse surgery
- 2 (Active Comparator): Group II, Prolapse repair and TVT 3 months afterwards if necessary
  Interventions: Procedure: Vaginal Repair for prolapse, TVT procedure; Procedure: TVT and Prolapse surgery

INTERVENTIONS:
Procedure: Vaginal Repair for prolapse, TVT procedure — 1. TVT at the time of Vaginal Repair
  2. TVT 3 months after Vaginal Repair
  Other Names: Incontinence surgery; Mid-urethra sling; Prolapse surgery.; Prolapse repair
Procedure: TVT and Prolapse surgery — 1. TVT at the time of Prolapse surgery
  2. TVT 3 months after Prolapse Surgery

SUMMARY:
It is unknown whether it is best to do the TVT( procedure for urinary stress incontinence in women) at the time of prolapse surgery or at a later date. Women with both conditions were randomized to both procedures together or the TVT 3 months after the prolapse surgery. Any or no leakage when couching was the main end-point, evaluated 1 year after the last surgery

DETAILED DESCRIPTION:
All women were evaluated by the POP-Q (pelvic Organ Prolapse Quantification) prior to surgery and 1 year after.

Examination for urinary leakage was done prior to surgery and 1 year after. Group 2 was also examined after prolapse surgery to see if TVT was still needed.

ELIGIBILITY:
Inclusion Criteria: Pelvic Organ Prolapse that needs surgical repair and objectively proven urinary stress incontinence -

Exclusion Criteria: Not agreed to participate in randomization

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2002-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Any or no leakage of urine when coughing | 1 year

SECONDARY OUTCOMES:
The cure of urinary stress incontinence (USI) by only prolapse surgery | 1 year
Result of prolapse surgery in two intervention strategies in women suffering from both genital prolapse and USI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Borstad, MD, Principal Investigator — Michael Abdelnoor Phd, Department of epidemiology (same hospital)